CLINICAL TRIAL: NCT07131579
Title: Regional Intravenous Analgesic Effect of Dexmedetomidine in Knee Surgeries Under Spinal Anesthesia: A Prospective, Randomized, Double-Blind Controlled Study
Brief Title: Intravenous Regional Analgesia of Dexmedetomidine
Acronym: Dexmedetomidin
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dexmedetomidine IV analgesia
Record Dates: First submitted 2025-08-06; First posted 2025-08-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Dexmedetomidine Analgesia; Knee Surgery
MeSH Terms: interventions — Saline Solution; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The patient will be allocated into one of two equal (1:1) groups according to the drug injected intravenously below the Pneumatic tourniquet after its inflation. Group D (Dexmedetomidine) will receive 0.5 mcg/kg of dexmedetomidine, diluted in normal saline while, group P (placebo) will receive same volume normal saline
Who Masked: Participant, Investigator
Masking Description: An anesthetist, not involved in the study , was responsible for randomization list construction, in blocks, opening the sealed envelopes and so, the preparation of the study drug
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): after spinal anesthesia; patient will receive normal saline injected intravenously below the Pneumatic tourniquet after its inflation
  Interventions: Drug: Normal Saline
- Dexmedetomidine (Active Comparator): after spinal anesthesia; patient will receive 0.5 mcg/kg dexmedetomidine, diluted in a normal saline injected intravenously below the Pneumatic tourniquet after its inflation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Normal Saline — equal volume of normal saline
  Arms: control
Drug: Dexmedetomidine — 0.5 mcg/kg of dexmedetomidine
  Arms: Dexmedetomidine

SUMMARY:
Dexmedetomidine is a highly selective α₂-adrenergic receptor agonist that exerts its effects by inhibiting the release of norepinephrine at presynaptic nerve terminals, leading to reduced sympathetic activity; This mechanism results in analgesia, sedation, and anxiolysis without significant respiratory depression

DETAILED DESCRIPTION:
In the context of intravenous regional anesthesia (IVRA), dexmedetomidine has been employed as an adjuvant to local anesthetics like lidocaine to improve block characteristics; Clinical studies have demonstrated that adding dexmedetomidine to lidocaine in IVRA accelerates the onset of sensory and motor blocks, extends the duration of postoperative analgesia, and reduces the incidence of tourniquet pain

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* American Society of Anesthesiologists (ASA) Physical Status Classification System I or II
* Scheduled for elective knee surgery under spinal anesthesia
* Body mass index (BMI) 18-30 kg/m²
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Hypersensitivity to dexmedetomidine
* Chronic kidney diseases serum creatinine >1.5 mg\dl or Patient has known renal disease
* Chronic opioid or sedative use
* Any cardiac conduction abnormalities
* Uncontrolled arterial hypertension
* Neuropathy
* Diabetes mellitus
* Impaired perfusion of the operative limb (Edema, Peripheral vascular Disease e.g "Raynaud Phenomenon")
* History or recent lower limb deep venous thrombosis (DVT) or Phlebitis
* Infection or vascular access limitation in the operated lower limbs
* Any contraindication of spinal anesthesia e.g "Coagulopathy"
* Any contraindications for tourniquet e.g "sickle cell anemia"

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
postoperative duration of analgesia | within 24 hours after the surgery
  the time measured from the study drug injection to the first request of analgesia by the patient

SECONDARY OUTCOMES:
total postoperative analgesic consumption | in the first 24-hour postoperative
  mg
Sedation levels | done Perioperatively at the following time points (Immediately before spinal anesthesia and immediately before tourniquet deflation. Then 5, 15, 30 min besides, 1, 2, 4, and 6 hours after tourniquet deflation)
  Ramsay Sedation Score (RSS) (the score from 1-6; where 1 = anxious, agitated, 2 =cooperatives, oriented, 3 =respond to command only, 4 =brisk response to stimulus, 5 =sluggish response to stimulus, 6 =no response to stimulus)
The time of sensory block regression in both lower limbs | Postoperatively every 15 min till full regression of the sensory block (score =0)
  using three-point scale via pinprick test over the limb in both limbs separately (where; 0 = Normal sensation (absent sensory block), 1 = Dull sensation (partial sensory block) and 2 = No sensation (complete sensory block)
The motor block regression time in both lower limbs | every 15 min till confirmation of full regression of the motor block (Modified Bromage Scale=0)
  using Modified Bromage Scale (0-3)
heart rate (HR), | preoperative, immediately after inject both spinal anesthesia and study drug, then every 5 minutes for the first 30 minutes and then every 15 minutes till end of the surgery. also, record after tourniquet deflation 5, 15, 30 min beside 1, 2, 4, 6 hours
  beat per minute
systolic blood pressure (SBP) | preoperative, immediately after inject both spinal anesthesia and study drug, then every 5 minutes for the first 30 minutes and then every 15 minutes till end of the surgery. also, record after tourniquet deflation 5, 15, 30 min beside 1, 2, 4, 6 hours
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine-Mansoura University, Al Mansurah, Egypt